CLINICAL TRIAL: NCT06133621
Title: Thrombophilia Assessment and Pregnancy: Determination of Reference Values for dRVVT in Pregnant Women
Brief Title: Determination of Reference Values for Diluted Russell's Viper Venom Time (dRVVT) Specific to Pregnant Women (GRAPL)
Acronym: GRAPL
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1016
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Normal Pregnancy
Keywords: Pregnancy; Thrombophilia; Antiphospholipid syndrome; Vascular diseases of pregnancy; Diluted Russell viper venom time
MeSH Terms: conditions — Thrombophilia; Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: Patients treated at HCL who have had an increased dRVVT ratio during pregnancy, investigated in the context of the development of VDP during pregnancy
  Interventions: Other: dosage dRVVT
- Controls: Patients with normal pregnancies followed at the Croix Rousse maternity hospital
  Interventions: Other: dosage dRVVT

INTERVENTIONS:
Other: dosage dRVVT — Blood test dRVVT assay on two tubes of blood in the haemostasis laboratory of the Center de Biologie et de Pathologie Est

SUMMARY:
Pregnancy is associated with significant changes in several aspects of haemostasis, especially an imbalance between procoagulant and anticoagulant factors. These changes contribute to creating a state of hypercoagulability, mainly at the end of pregnancy and during the post-partum period, protecting pregnant women from delivery haemorrhage, but exposing them to a major thromboembolic risk.

Vascular diseases of pregnancy (VDP) are obstetric diseases which are linked to an ischaemic origin associated with placental thrombosis. These include pre-eclampsia, retroplacental haematoma, intrauterine growth retardation and even foetal death in utero. A number of risk factors have been identified for these VDPs, some of which have extremely serious consequences, the main one being antiphospholipid syndrome (APS).

The diagnosis of VDP in a current or previous pregnancy requires close monitoring and joint management by an obstetrician, haemostasis physician, internist and medical biologist, particularly in terms of pre, peri- and post-partum anticoagulation in patients at increased risk of thromboembolism.

The aim of treating APS during pregnancy is : to reduce the occurrence of maternal arterial or venous thrombotic complications in one hand and in the other hand to reduce the occurrence of obstetric complications, which are responsible of a significant morbimortality rate. The detection of a possible APS during pregnancy will therefore determine the specific management of patients.

The latest guidelines from the Groupe Français d'Etude sur l'Hémostase et la Thrombose (GFHT) in 2022 recommended a diluted Russell's viper venom time (dRVVT) and an activated partial thromboplastin time (APTT) measured using a sensitive reagent such as silica (SCT) should be used to assess the presence of LA.

DETAILED DESCRIPTION:
Please remove all personal pronouns. For example, please change "we" to "the investigators" and "you" to "participants." The "Control + Find" function (Ctrl+F) can be used to locate personal pronouns throughout the record.

ELIGIBILITY:
Inclusion Criteria:

Control group :

* patients with normal pregnancies at the HCL.
* Affiliation to a social security regime

Case group :

* Patients followed at the HCL who had an increased dRVVT ratio during pregnancy, investigated as part of the development of VDP during pregnancy.
* Affiliation to a social security regime

Exclusion Criteria:

* History of thromboembolic disease
* History of autoimmune disease
* History of VDP

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Selection by the gynaecologist of pregnant women at the Croix Rousse maternity hospital, who presenting a physiological pregnancy with no history of thromboembolic or autoimmune pathology or vascular disease of pregnancy
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-09-28 (Actual); Study Completion 2025-09-28 (Actual)

PRIMARY OUTCOMES:
dRVVT value during pregnancy. | through study completion, an average of 9 months
  Carrying out the dRVVT in the haemostasis laboratory of the Centre de Biologie et de Pathologie Est

CONTACTS AND LOCATIONS:
Overall Officials: Céline DR BAZIN, DR, Principal Investigator — Laboratoire d'hémostase CBPE HCL
Locations (1):
- Dr Céline BAZIN, Lyon, France